CLINICAL TRIAL: NCT05198011
Title: Mandibular Ridge Augmentation Using Three-Dimensional Printed Model for Customization of Titanium Mesh
Brief Title: Three-Dimensional Printed Customized Titanium Mesh for Mandibular Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Augmentation_Maxillo
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D mandibular ridge augmentation (Experimental)
  Interventions: Procedure: 3D customized Titanium Mesh (Study)
- Conventional mandibular ridge augmentation (Active Comparator)
  Interventions: Procedure: Conventional ridge augmentation (Control)

INTERVENTIONS:
Procedure: 3D customized Titanium Mesh (Study) — approach for planning and augmenting atrophic posterior mandibular ridge using a pre-customized TiMe on a 3D model. The 3D surgical model will be virtually created from a cone-beam computed tomography (CBCT) and printed using Fused deposition modeling (FDM) machine. The 3D model will be then used to contour the TiMe in accordance with the needed amount of augmentation then will be used to help pack and contour the graft material.
  Arms: 3D mandibular ridge augmentation
Procedure: Conventional ridge augmentation (Control) — the conventional technique of ridge augmentation using Titanium Mesh
  Arms: Conventional mandibular ridge augmentation

SUMMARY:
Completely or partially edentulous patients suffer from resorption of the alveolar bone, they always seek rehabilitation which becomes challenging. Alveolar ridge augmentation is widely done now to offer these patients functional and esthetic restoration. Many techniques have been proposed to obtain good results of ridge augmentation. Titanium Mesh (TiMe) is widely used, also digital and computer-guided surgery now plays an important role to improve the techniques and results in ridge augmentation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have a posterior mandibular atrophic ridge
* Distance between the crest of the ridge and the superior border of the inferior alveolar canal will be from 5 mm to 7 m
* Adequate inter-arch space

Exclusion Criteria:

* Patients who have any uncontrolled systemic disease contraindicated to oral surgery ( Diabetes, hypertension, and patients under chemotherapy treatment )
* Patients who have any relevant bone disease.
* Patients who are smokers

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in bone volume | at baseline and 6 months
  Bone volume wa measured using CBCT
Operation time | During the procedure
  Time of operation for each group will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt